CLINICAL TRIAL: NCT05201703
Title: Pilot Study of Add-On Fycompa (Perampanel)Treatment for Catamenial Epilepsy
Brief Title: Fycompa in Catamenial Epilepsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Florida (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202102694
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Catamenial Epilepsy
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fycompa 4 mg daily (Experimental)
  Interventions: Drug: Fycompa
- Fycompa 4 mg daily with a boost to 6 mg daily (Active Comparator)
  Interventions: Drug: Fycompa with a boost

INTERVENTIONS:
Drug: Fycompa — Fycompa 4 mg daily
  Other Names: Perampanel
  Arms: Fycompa 4 mg daily
Drug: Fycompa with a boost — Fycompa 4 mg daily with a boost to 6 mg daily a week before the start of your menstruation cycle until Day 4 of your cycle.
  Other Names: Perampanel
  Arms: Fycompa 4 mg daily with a boost to 6 mg daily

SUMMARY:
The purpose of the proposed investigation is to carry out a pilot study of add-on perampanel (Fycompa) in women with perimenstural (C1) catamenial epilepsy. Perampanel, a noncompetitive AMPA receptor antagonist, is uniquely positioned to decrease progesterone receptor mediated excitotoxicity. This mechanism of action would allow a novel use of perampanel as an effective treatment of C1 catamenial epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of focal onset seizures (FOS) i. Established by clinical history and an EEG ii. Patients with a normal EEG may be included if they met other diagnostic criteria based on clinical history
* Presumably ovulatory women based on menstrual cycles of 21-35 days from beginning of menstrual flow to the beginning of the next menses
* ≥18-50 years old
* ≥2 unprovoked seizures per month despite drug trials with ≥1 first-line anti-epileptic drugs (AED)
* Seizures must show a C1 catamenial pattern in 2 of 3 documented cycles i. C1 pattern will be defined as a two-fold increase in average daily seizure frequency during the menstrual phase, as compared to the follicular and luteal phases of the ovulation cycle, in 2 of 3 documented cycles. The menstrual phase will be defined as days -3 to +3 of the menstrual cycle (where onset of menstruation is defined as day 1) (Herzog et al, 1997). Of note, in the NIH Progesterone Trial, the level of catameniality was 1.69 based on Herzog et al. (1997) criteria though this trial will use a level of 2 to include women only with high levels of perimenstrual catamenial exacerbation.
* Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

* Progressive neurologic or systemic disorder
* Use of systemic hormonal contraception during 3 months prior to enrollment (however, subjects with a progestin-releasing IUD who still have monthly periods may be enrolled)

  a. Women on system hormonal contraception will be excluded as these women are not ovulatory
* Subject is pregnant or breastfeeding
* Active suicidal or homicidal ideation
* Comatose individuals.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study is enrolling women of child bearing potential to investigate the use of perampanel in women with perimenstrual catamenial epilepsy
Enrollment: 7 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Zarroli, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * 1 subject was excluded from the study due to a positive C-SSRS.
  * 2 subjects were excluded during the baseline period (1 subject did not have her menstrual period during the baseline period so dropped out due to irregular menses and 1 subject did not have any seizures during the baseline phase).
Period: Overall Study
Arm/Group | Fycompa 4 mg Daily | Fycompa 4 mg Daily With a Boost to 6 mg Daily
Started | 1 | 3
Completed | 1 | 1
Not Completed | 0 | 2
Not completed — Did not understand how to boost medication despite counseling; did not boost | 0 | 1
Not completed — Subject did not tolerate the treatment (perampanel) due to mild side effects so exited the study. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fycompa 4 mg Daily | Fycompa 4 mg Daily With a Boost to 6 mg Daily | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 36.5 [33 to 40] | 31.7 [25 to 39] | 33.6 [25 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate (Percent of Patients Experiencing a 50% or Greater Reduction in Seizures) Relative to Baseline Seizure Frequencies
Description: To measure the 50% responder rate will be analyzed using Chi square analysis.
Time Frame: Baseline (2 months) and treatment (2 months)
Population: Statistics unable to be performed due to low sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | Fycompa 4 mg Daily | Fycompa 4 mg Daily With a Boost to 6 mg Daily
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 4 months per participant assessment (2 months of baseline and 2 months of treatment)
Arm/Group | Fycompa 4 mg Daily | Fycompa 4 mg Daily With a Boost to 6 mg Daily
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fycompa 4 mg Daily (N=1) | Fycompa 4 mg Daily With a Boost to 6 mg Daily (N=3)
Feeling off (Nervous system disorders) | 0 (0) | 1 (1) — Patient just felt "off" and not like herself on medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05201703/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05201703/SAP_002.pdf